CLINICAL TRIAL: NCT01740206
Title: Should Chronic Stimulant Medications be Continued Preoperatively in Patients With Attention Deficit Hyperactivity Disorder(ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Richard Cartabuke, Co-Director of Outpatient Anesthesia Services, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00721
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amphetamine and/or methylphenidate (Active Comparator): Patients who took their amphetamine and/or methylphenidate the morning of surgery.
  Interventions: Drug: Amphetamine and/or methylphenidate
- Hold stimulant medication (Experimental): Patients who did not take their stimulant medication the morning of surgery.
  Interventions: Other: Hold stimulant medication

INTERVENTIONS:
Drug: Amphetamine and/or methylphenidate — Patients who took their stimulant medication the day of surgery.
  Arms: Amphetamine and/or methylphenidate
Other: Hold stimulant medication — Patients who held their stimulant medication the day of surgery.
  Arms: Hold stimulant medication

SUMMARY:
Patients on chronic stimulant therapy for the treatment of Attention deficit hyperactivity disorder (ADHD) who are undergoing an outpatient surgical or diagnostic procedure will be randomized to one of two groups: stimulant medication administered on the day of surgery or stimulant medication withheld on the day of surgery. The choice of anesthetic pharmacology will be at the discretion of the attending anesthesiologist, but the endpoint will be a bispectral index (BIS) between 40 and 60 to ensure adequate and similar depth of anesthesia. Blood pressure, heart rate and use of vasopressors or anticholinergics will be recorded and the incidence of hypotension, bradycardia, or administration of medications will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled if they have been diagnosed with ADHD and have been taking amphetamines and/or methylphenidate for at least the last six months and are undergoing an outpatient surgical or diagnostic procedure.

Exclusion Criteria:

* Patients will be excluded if they are taking antidepressant medications, anxiolytic medication, analgesia medications other than acetaminophen or NSAIDs, if they have an allergy to midazolam, or a have cardiac disease.
* Procedures that entail the likelihood of blood transfusion will be excluded.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects with unknown ADHD medication status were excluded from the analysis.
Groups:
- Patients Taking ADHD Medication: Patients who took their amphetamine and/or methylphenidate the morning of surgery.
- Patients Not Taking ADHD Medication: Patients who held their stimulant medication the day of surgery.
Period: Overall Study
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Started | 14 | 34
Completed | 14 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication | Total
Number analyzed (Participants) | 14 | 34 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.25 (2.56) | 9.35 (2.79) | 9.32 (2.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 11 | 23 | 34

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Heart rate prior to anesthetic induction
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 14 | 34
BPM | 96.7 (13.9) | 88 (14)

2. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure prior to anesthetic induction
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 14 | 34
mmHg | 113.6 (13.5) | 109.2 (12.4)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure prior to anesthetic induction
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 14 | 34
mmHg | 71.1 (11) | 67.9 (9.3)

4. Secondary Outcome: Mean Blood Pressure
Description: Mean blood pressure prior to anesthetic induction
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 14 | 34
mmHg | 85.3 (10.5) | 81.7 (8.6)

5. Secondary Outcome: mYPAS Measurement in Patients Receiving Midazolam
Description: modified Yale Preoperative Anxiety Scale (mYPAS), which is commonly used for assessing anxiety during the induction of anesthesia, administered to patients who received midazolam prior to anesthesia induction.
  Assessment items: Activity (A) 1-4 points (A = score/4), Vocalizations (V) 1-6 points (V = score/6), Emotional expressivity (E) 1-4 points (E = score/4), State of arousal (S) 1-4 points (S = score/4), Use of parent (U) 1-4 points (U = score/4). Final score = [(A + V + E + S +U)/5] x 100. Higher score = more anxiety.
Time Frame: Day 1
Population: Of the 48 subjects analyzed, 10 subjects received midazolam prior to their surgical procedure.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 4 | 6
scores on a scale | 30 [26 to 33] | 26 [23 to 42]

6. Secondary Outcome: mYPAS Measurement in Patients Not Receiving Midazolam
Description: modified Yale Preoperative Anxiety Scale (mYPAS), which is commonly used for assessing anxiety during the induction of anesthesia, administered to patients who did not receive midazolam prior to anesthesia induction.
  Assessment items: Activity (A) 1-4 points (A = score/4), Vocalizations (V) 1-6 points (V = score/6), Emotional expressivity (E) 1-4 points (E = score/4), State of arousal (S) 1-4 points (S = score/4), Use of parent (U) 1-4 points (U = score/4). Final score = [(A + V + E + S +U)/5] x 100. Higher score = more anxiety.
Time Frame: Day 1
Population: Of the 48 subjects analyzed, 38 subjects did not receive midazolam prior to their surgical procedure.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Number analyzed (Participants) | 10 | 28
scores on a scale | 28 [23 to 42] | 28 [23 to 28]

ADVERSE EVENTS:
Arm/Group | Patients Taking ADHD Medication | Patients Not Taking ADHD Medication
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/34
Other Adverse Events (participants affected / at risk) | 0/14 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes